CLINICAL TRIAL: NCT06081738
Title: Evaluation of The Effects of Neostigmine Versus Sugammadex on Renal Functions in Laparoscopic Cholecystecomy A Randomized Controlled Study
Brief Title: Neostigmine Versus Sugammadex on Renal Functions
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2/2023ANSTH49
Record Dates: First submitted 2023-09-23; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Sugammadex; Neostigmine
MeSH Terms: interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neostigmine Group (Active Comparator)
  Interventions: Drug: Neostigmine
- Sugammadex Group (Active Comparator)
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — a combination of 0.04 mg/kg neostigmine with 0.01 mg/kg atropine intravenously at the reappearance of a second twitch of TOF after the last dose of rocuronium
  Arms: Neostigmine Group
Drug: Sugammadex — 2-4 mg/kg sugammadex intravenously upon the reappearance of a post-tetanic count 1-2 or a second twitch of TOF after the last dose of rocuronium
  Arms: Sugammadex Group

SUMMARY:
The study will assess the acute effects of sugammadex or neostigmine on renal function as determined with more specific and sensitive tests in laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

* normal renal function (serum Cr 0.4- 1.4 g/dL)
* American Society of Anesthesiologists (ASA) Class I-II

Exclusion Criteria:

* Incapacity to consent.
* Pre-existing impaired kidney functions.
* Severe neuromuscular disease, as: myasthenia gravis & muscular dystrophy.
* Intra-operative bleeding
* Lengthy operations that exceed 2 hours.
* Hemodynamic changes more than 20% of the base line

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
neutrophil gelatinase associated lipocalin (NGAL) values | baseline ( 2 days preoperative) and 12 hours after surgery
  normal overall unisex value 47-55 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No